CLINICAL TRIAL: NCT00307619
Title: Randomized, Double-blind Placebo Controlled Trial With Topiramate for the Treatment of Obese Patients With Binge Eating Disorder
Brief Title: An Efficacy and Tolerability Study for Topiramate in Obese Patients With Binge Eating Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003667
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Binge Eating
Keywords: Binge-Eating Disorder
MeSH Terms: conditions — Bulimia; Binge-Eating Disorder | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the effectiveness and tolerability of topiramate compared to placebo in patients with binge eating disorder receiving Cognitive Behavior Therapy (CBT)

DETAILED DESCRIPTION:
This was a 21-week multicenter, double-blind, parallel-group, randomized controlled trial comparing the efficacy and tolerability of an add-on treatment with 200mg of topiramate versus placebo in obese patients with BED receiving group CBT. The aim of this trial is to investigate the efficacy and tolerability of adjunctive topiramate to CBT in obese patients with BED through improvement in binge eating, related psychopathology, and weight loss. The study hypothesis is that the patients using topiramate + CBT will loose more weight than patients using placebo + CBT.Tolerability will be investigated through reported adverse events and dropouts, with reasons for leaving the study being analyzed. The randomized patients will receive capsules of topiramate (25 mg, 50 mg) or placebo correspondent daily for 21 weeks

ELIGIBILITY:
Inclusion Criteria:

* Have been meeting the diagnostic criteria for binge eating disorder (according to the Diagnostic and Statistical Manual for Mental Disorders - IV Edition criteria) with at least 2 days of binge eating per week and severity at least moderate defined by binge eating scale (score = 17)
* BMI = > 30 kg/m2 to < 46 kg/m2
* Women must be post menopausal for at least one year or surgically sterilized (hysterectomy, tubal ligation), or practice sexual abstinence or use an acceptable method of birth control (i.e. a hormonal contraceptive, spermicide plus barrier method, intrauterine device and/or vasectomized partner)

Exclusion Criteria:

* Has a history or actual diagnostic of significant psychiatric disorder (schizophrenia, psychosis, major affective disorder, suicide risk, dementia, abuses alcohol or other drugs)
* has a malignancy or a history of malignancy within the past 5 years (except basal cell carcinoma)
* evidence of uncontrolled thyroid disorders
* uncontrolled hypertension (defined as a diastolic blood pressure >110 mm/Hg and/or a systolic blood pressure >180 mm/Hg with or without medication). Hypertensive patients on medications must have been on the same dose of the same antihypertensive medication for at least two months
* history or significant renal failure or glaucoma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2003-11; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Weight, Body Mass Index,number of binge eating and anthropometric measurements

SECONDARY OUTCOMES:
changes in blood pressure, serum triglycerides levels, serum cholesterol levels, beck depression scale scores.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.

REFERENCES:
- [Derived] Claudino AM, de Oliveira IR, Appolinario JC, Cordas TA, Duchesne M, Sichieri R, Bacaltchuk J. Double-blind, randomized, placebo-controlled trial of topiramate plus cognitive-behavior therapy in binge-eating disorder. J Clin Psychiatry. 2007 Sep;68(9):1324-32. doi: 10.4088/jcp.v68n0901. PMID 17915969